CLINICAL TRIAL: NCT06800274
Title: A Randomized, Single-Blind Clinical Investigation to Compare the Efficacy and Safety of N-Acetyl-Aspartyl-Glutamate (NAAGA) Versus Azelastine Eye Drops in Patients With Allergic Conjunctivitis Associated With Tear Film Dysfunction
Brief Title: Clinical and Biological Evaluation of NAAGA Versus Azelastine Eye Drops in Allergic Subjects With Tear Film Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other)
Responsible Party: Principal Investigator, Mario Troisi, MD, Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASL Napoli 3 sud n. 31/2019
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Allergic Conjunctivitis; Dry Eye Disease (DED)
Keywords: allergic conjunctivitis; dry eye disease (DED); tear film dysfunction; azelastine; antihistamine eye drops; N acetyl-aspartyl glutamic acid (NAAGA)
MeSH Terms: conditions — Conjunctivitis, Allergic; Dry Eye Syndromes | interventions — isospaglumic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAAGA Group (Experimental)
  Interventions: Drug: NAAGA (N-acetyl-aspartyl-glutamate) 49 mg/mL
- Azelastine Group (Active Comparator)
  Interventions: Drug: azelastine hydrochloride 0.05%

INTERVENTIONS:
Drug: NAAGA (N-acetyl-aspartyl-glutamate) 49 mg/mL — 80 patients were randomly assigned to NAAGA in single dose (49 mg/mL), instilled as 1 drop per eye four times daily for four weeks. Specific diagnostic tests and procedures for dry eye disease were performed at week 0 (baseline), week 2 and week 4.
  Arms: NAAGA Group
Drug: azelastine hydrochloride 0.05% — 54 patients were randomly assigned to azelastine hydrochloride 0.05% instilled as 1 drop per eye 2 times a day in the conjunctival sac for for four weeks. Specific diagnostic tests and procedures for dry eye disease were performed at week 0 (baseline), week 2 and week 4.
  Arms: Azelastine Group

SUMMARY:
This randomized, single-blind study aims to compare the efficacy and safety of N-acetyl-aspartyl-glutamate (NAAGA) and azelastine hydrochloride eye drops in patients with allergic conjunctivitis associated with tear film dysfunction. A total of 134 atopic patients with mild-to-moderate tear film dysfunction were included. Participants were randomly assigned to receive either NAAGA (49 mg/mL, four times daily) or azelastine (0.05%, twice daily) for four weeks. The primary endpoint is the change in Ocular Surface Disease Index (OSDI) scores from baseline to week 4. Secondary endpoints include tear osmolarity, Schirmer test results, tear break-up time (TBUT), MMP-9 levels, and corneal staining scores. This study seeks to provide evidence for the tailored management of allergic conjunctivitis and tear film dysfunction.

DETAILED DESCRIPTION:
There is limited but growing evidence in the literature regarding the effectiveness of N-acetyl-aspartyl-glutamate (NAAGA) in managing allergic conjunctivitis, particularly in patients with concomitant tear film dysfunction. NAAGA is a neuropeptide with dual activity as a mast cell stabilizer and anti-inflammatory agent, reducing histamine release and mitigating inflammatory cascades such as leukotriene production and complement activation. These mechanisms address both the allergic and inflammatory components of ocular surface diseases. Despite its promising therapeutic potential, studies directly comparing NAAGA to other treatments, particularly H1 receptor antagonists like azelastine, remain scarce.

In previous studies, NAAGA has demonstrated efficacy in reducing ocular surface inflammation, improving tear film stability, and alleviating symptoms of dry eye disease (DED). It has been reported a significant reduction in inflammatory markers, such as HLA-DR expression, and improvement in tear break-up time (TBUT) and Ocular Surface Disease Index (OSDI) scores in patients treated with NAAGA. Another investigation comparing NAAGA to cyclosporine A noted faster symptom relief and fewer adverse effects with NAAGA, highlighting its tolerability and potential for broader application. However, the literature lacks robust, head-to-head comparisons of NAAGA with second-generation antihistamines, such as azelastine, in the context of allergic conjunctivitis with tear film dysfunction.

Based on this background, this randomized, single-blind trial is designed to compare the efficacy and safety of NAAGA (49 mg/mL) with azelastine hydrochloride (0.05%) in treating patients with mild-to-moderate allergic conjunctivitis associated with tear film dysfunction. Both treatments target key mechanisms of disease but differ in their primary mode of action. NAAGA offers dual anti-inflammatory and mast cell-stabilizing effects, while azelastine acts predominantly as an H1 receptor antagonist with additional mast cell stabilization.

The primary objective of this study is to demonstrate that NAAGA is non-inferior to azelastine in improving symptoms and clinical parameters of allergic conjunctivitis associated with tear film dysfunction. Specifically, the study will evaluate changes in the Ocular Surface Disease Index (OSDI) score over four weeks of treatment. Secondary objectives include assessing changes in tear osmolarity, TBUT, Schirmer test results, MMP-9 levels, and corneal staining scores, as well as patient-reported symptoms of ocular discomfort.

This trial will include 134 patients with atopy and mild-to-moderate tear film dysfunction, randomized to receive either NAAGA eye drops (administered four times daily) or azelastine eye drops (administered twice daily) for four weeks. Both groups will undergo comprehensive evaluations, including the OSDI questionnaire, tear osmolarity testing, Schirmer I test, TBUT measurement, MMP-9 assessment, and fluorescein staining of the ocular surface. Patient-reported discomfort will be tracked through weekly diaries.

The investigation is expected to provide critical insights into the comparative efficacy and safety of NAAGA and azelastine in this patient population. NAAGA's dual-action profile may offer broader therapeutic benefits, particularly in addressing inflammation-driven tear film instability and ocular surface damage. Results from this study could inform clinical decision-making and support the development of more targeted, personalized treatments for patients with allergic conjunctivitis and tear film dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with atopy confirmed by skin prick tests, elevated specific IgE levels, or Prist result >100 kU/L.
* Mild-to-moderate tear film dysfunction defined by OSDI scores ≥13 and at least one diagnostic abnormality (TBUT <10 sec, Schirmer I test <10 mm, CLEK score for corneal staining >1, or tear osmolarity >308 mOsm/L).

Exclusion Criteria:

* Severe ocular surface disorders
* Unilateral dry eye syndrome.
* Recent ocular surgery (within 3 months) or refractive surgery (within 6 months).

  . - Active ocular infections.
* Previous herpetic keratitis.
* Systemic or topic therapies with steroids in the last three months.
* Local therapies in the last 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Improvement in Ocular Surface Disease Index (OSDI) Score from Baseline | Week 4
  The OSDI is a validated questionnaire used to measure the severity of dry eye disease and its impact on vision-related quality of life. It includes 12 questions divided into three subscales: ocular symptoms, vision-related functions, and environmental triggers. Each item is scored on a scale from 0 ("none of the time") to 4 ("all of the time"). The total OSDI score is calculated on a scale of 0 to 100, with higher scores indicating greater severity. A clinically meaningful change is defined as a decrease of ≥10 points.

SECONDARY OUTCOMES:
Improvement in OSDI Score from Baseline | Week 2
  The OSDI score, as described above, will also be evaluated at an intermediate time point to track early symptom relief. The total OSDI score is calculated on a scale of 0 to 100, with higher scores indicating greater severity. A clinically meaningful change is defined as a decrease of ≥10 points.
Changes in Tear Osmolarity from Baseline | Week 2 and Week 4
  Tear osmolarity will be measured using a TearLab osmometer. Tear samples will be collected from the inferior tear meniscus, and osmolarity will be expressed in mOsm/L. Elevated tear osmolarity (>308 mOsm/L) is a hallmark of dry eye disease. A reduction in tear osmolarity reflects improved tear film stability and reduced ocular surface stress.
Improvement in Tear Break-Up Time (TBUT) from Baseline | Week 2 and Week 4
  The TBUT will be measured using fluorescein dye and a cobalt-blue filtered slit lamp. The time from the last blink to the first visible break in the tear film will be recorded in seconds. Two readings will be averaged unless they differ by more than 2 seconds, in which case a third reading will be included. TBUT values of less than 10 seconds indicate tear film instability.
Improvement in Schirmer's Test 1 Results from Baseline | Week 2 and Week 4
  The Schirmer's test will measure total tear production, including both basal and reflex tearing. A 35 mm x 5 mm strip of filter paper will be placed in the lower conjunctival sac for 5 minutes. The length of wetting in millimeters will be recorded. A normal value is considered >10 mm in 5 minutes, while dry eye is diagnosed at <5 mm.
Reduction in MMP-9 Positivity from Baseline | Week 4
  Inflammation will be assessed using the InflammaDry® test to detect matrix metalloproteinase-9 (MMP-9) levels in tear fluid. MMP-9 is an inflammatory marker elevated in dry eye disease. Results will be reported as positive or negative.
Improvement in Corneal Staining Scores | Week 4
  Corneal staining will be evaluated using fluorescein dye and the National Eye Institute (NEI)/Industry Workshop guidelines. The cornea will be divided into five regions (central, superior, inferior, nasal, and temporal), with each region graded on a 0-3 scale, yielding a total score of 0-15. Higher scores indicate more severe staining and damage.
Patient-Reported Changes in Ocular Discomfort | Week 4
  Participants will maintain weekly symptom diaries to report ocular discomfort. Scores will be evaluated on a 5-point Likert scale, with higher scores indicating greater symptom severity.
Incidence of Treatment-Emergent Adverse Events (TEAEs) | Week 4
  Safety and tolerability will be assessed by recording the incidence and nature of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse device effects (ADEs), and serious ADEs (SADEs) throughout the study. Investigational Medical Device Deficiencies (IMDDs) will also be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Troisi, MD, Principal Investigator — Azienda Ospedaliera Universitaria OO.RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno, Italy
Locations (1):
- Azienda Ospedaliera Universitaria OO.RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno, Salerno, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Suarez-Cortes T, Merino-Inda N, Benitez-Del-Castillo JM. Tear and ocular surface disease biomarkers: A diagnostic and clinical perspective for ocular allergies and dry eye disease. Exp Eye Res. 2022 Aug;221:109121. doi: 10.1016/j.exer.2022.109121. Epub 2022 May 21. PMID 35605673
- [Background] Shin D, Sang Min J. Comparison of treatment effects between 4.9% N-acetyl-aspartyl glutamic acid and 0.05% cyclosporine A eye drops in dry eye patients. Graefes Arch Clin Exp Ophthalmol. 2022 Oct;260(10):3285-3291. doi: 10.1007/s00417-022-05682-x. Epub 2022 Apr 29. PMID 35486175
- [Background] Regu VR, Swain RP, Subudhi BB. Drug Delivery for Ocular Allergy: Current Formulation Design Strategies and Future Perspectives. Curr Pharm Des. 2023;29(33):2626-2639. doi: 10.2174/0113816128275375231030115828. PMID 37936454
- [Background] Leonardi A, Quintieri L, Presa IJ, LLoves JM, Montero J, Benitez-Del-Castillo JM, Leston FJS, Gonzalez-Mancebo E, Asero R, Groblewska A, Kuna P. Allergic Conjunctivitis Management: Update on Ophthalmic Solutions. Curr Allergy Asthma Rep. 2024 Jul;24(7):347-360. doi: 10.1007/s11882-024-01150-0. Epub 2024 Jun 13. PMID 38869807
- [Background] Kumar N, Feuer W, Lanza NL, Galor A. Seasonal Variation in Dry Eye. Ophthalmology. 2015 Aug;122(8):1727-9. doi: 10.1016/j.ophtha.2015.02.013. Epub 2015 Apr 6. No abstract available. PMID 25912217
- [Background] Janeczko P, Norris MR, Bielory L. Assessment of receptor affinities of ophthalmic and systemic agents in dry eye disease. Curr Opin Allergy Clin Immunol. 2021 Oct 1;21(5):480-485. doi: 10.1097/ACI.0000000000000773. PMID 34387278
- [Background] James IG, Campbell LM, Harrison JM, Fell PJ, Ellers-Lenz B, Petzold U. Comparison of the efficacy and tolerability of topically administered azelastine, sodium cromoglycate and placebo in the treatment of seasonal allergic conjunctivitis and rhino-conjunctivitis. Curr Med Res Opin. 2003;19(4):313-20. doi: 10.1185/030079903125001785. PMID 12841924
- [Background] Jambou D, Lapalus P. Effect of N-acetyl-aspartyl-glutamate (Naaga) on in-vitro leukotriene synthesis by macrophage cell line P388D1. Int J Tissue React. 1990;12(5):273-80. PMID 1983004
- [Background] Herrero-Vanrell R, Jauregui Presa I, Leceta Bilbao A, Montero-Iruzubieta J. Fundamental Aspects and Relevance of Components in Antihistamine Eye Drops. J Investig Allergol Clin Immunol. 2023 Dec;33(6):431-438. doi: 10.18176/jiaci.0963. PMID 38095492
- [Background] Goldschmidt PL, Vulliez-Le Normand B, Briquet I, Dray F. Effects of N-acetyl-aspartyl glutamic acid and sodium cromoglycate on leukotriene B4 secretion by human leukocytes. Allergy. 1990 Jul;45(5):363-9. doi: 10.1111/j.1398-9995.1990.tb00512.x. PMID 2165751
- [Background] Garcia-Queiruga J, Pena-Verdeal H, Sabucedo-Villamarin B, Garcia-Resua C, Giraldez MJ, Yebra-Pimentel E. Temporal Progression of Entry Factors into the Vicious Circle of Dry Eye in Untreated Sufferers. Life (Basel). 2024 Jun 26;14(7):806. doi: 10.3390/life14070806. PMID 39063561
- [Background] Fukuda K, Kishimoto T, Sumi T, Yamashiro K, Ebihara N. Biologics for allergy: therapeutic potential for ocular allergic diseases and adverse effects on the eye. Allergol Int. 2023 Apr;72(2):234-244. doi: 10.1016/j.alit.2022.09.005. Epub 2022 Nov 1. PMID 36333219
- [Background] El Fekih L, Khairallah M, Ben Amor H, Mahmoud A, Chiambaretta F, Messaoud R. Successful management of dry eye disease with a new eye drop formulation combining hyaluronic acid, trehalose, and N-acetyl-aspartyl-glutamic acid (NAAGA). J Fr Ophtalmol. 2024 Sep;47(7):104169. doi: 10.1016/j.jfo.2024.104169. Epub 2024 Jun 4. PMID 38838456